CLINICAL TRIAL: NCT01102686
Title: Proposed Investigator-Initiated Clinical Trial of Pyrimethamine as a Treatment for Late-Onset GM2-gangliosidosis (Tay-Sachs and Sandhoff Disease)
Brief Title: Pyrimethamine as a Treatment for Late-Onset GM2-gangliosidosis (Tay-Sachs and Sandhoff Disease)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1000013660
Record Dates: First submitted 2009-10-16; First posted 2010-04-13 (Estimated); Last update posted 2012-02-23 (Estimated); Status verified 2012-02

CONDITIONS: Gangliosidoses, GM2; Sandhoff Disease; Tay-Sachs Disease
Keywords: Late-onset GM2-gangliosidosis; pyrimethamine
MeSH Terms: conditions — Gangliosidoses, GM2; Sandhoff Disease; Tay-Sachs Disease | interventions — Pyrimethamine; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pyrimethamine (Experimental)
  Interventions: Drug: Pyrimethamine; Drug: Leucovorin

INTERVENTIONS:
Drug: Pyrimethamine — Pyrimethamine will be taken orally as a single daily dose of 25 mg/day for 4 weeks, then increasing by 25 mg per dose in three four-week steps, to a final dose of 100 mg/day
Drug: Leucovorin — To eliminate or minimize potential hematologic effects of Pyrimethamine, Leucovorin is to be co-administered with Pyrimethamine at a dose level of 5 mg per day, given when Pyrimethamine is administered.

SUMMARY:
The objectives of this clinical trial are to assess the safety and tolerability, as well as efficacy, of a stepwise dosing regimen of pyrimethamine, starting at 25 mg/day, given as a single dose daily for 4 weeks in patients affected with chronic Tay-Sachs or Sandhoff variants.

DETAILED DESCRIPTION:
Patients with late-onset Tay-Sachs or Sandhoff disease will be given increasing doses of Pyr, up to but not exceeding doses used to treat malaria, over a 5-month period. We will follow the effect of the treatment on the levels of Hex A enzyme activity in white blood cells, which are considered to be a reflection of the likely enzyme activity in the brain. We will also follow some other lysosomal enzyme activities to determine if the effect is specific for Hex A. Furthermore, we will examine the effect of the treatment on the levels of GM2-ganglioside in the white blood cells. On the basis of the studies done on cultured skin cells, we expect that treatment with Pyr will increase the levels of Hex A and decrease the accumulation of GM2-ganglioside in the white blood cells.

ELIGIBILITY:
Inclusion Criteria:

* biochemically and genetically confirmed diagnosis of GM2-gangliosidosis caused by β-hexosaminidase deficiency resulting from mutations in the HEXA or HEXB genes;
* having HEXA or HEXB mutations shown to be responsive to pyrimethamine in vitro;
* over 17 years of age at the time of study initiation;
* able to understand and cooperate with the requirements of the study protocol;
* mentally competent, have the ability to understand and willingness to sign the informed consent form;
* able to travel to one of the three participating study sites;
* women of child-bearing potential must use accepted contraceptive methods and must have a negative serum or urine pregnancy test within one week prior to treatment initiation;
* fertile men must practice effective contraceptive methods during the study period, unless documentation of infertility exists;
* laboratory values ≤2 weeks prior to randomization must show adequate hematologic, hepatic, renal, and coagulation function; and body weight >40 kg.

Exclusion Criteria:

* serious medical illness, significant cardiac disease or severe debilitating pulmonary disease;
* any hematologic abnormality, especially megaloblastic anemia, leukopenia, thrombocytopenia, pancytopenia;
* any active uncontrolled bleeding or any bleeding diathesis (e.g., active peptic ulcer disease);
* possible folate deficiency, and those receiving therapy (such as phenytoin) affecting folate levels;
* any complex disease that may confound treatment assessment;
* pregnant women or women of child-bearing potential not using reliable means of contraception;
* lactating females;
* fertile men unwilling to practice contraceptive methods during the study period;
* unwilling or unable to follow protocol requirements;
* known hypersensitivity reactions, intolerance or adverse reactions to pyrimethamine;
* evidence of active infection, or serious infection within the past month;
* HIV infection;
* a history of cancer of any type;
* receiving any other standard or investigational treatment for any indication within the past 4 weeks prior to initiation of pyrimethamine treatment;
* receiving immunotherapy of any type within the past 4 weeks prior to initiation of pyrimethamine treatment; or any condition or abnormality, which may, in the opinion of the investigator, compromise the safety of patients.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-08; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Efficacy of pyrimethamine | Baseline, before exposure to pyrimethamine, and Weeks 4, 8, 12, 16 and 18.
  Changes in Hex A and Hex B, β-glucuronidase using blood assays

SECONDARY OUTCOMES:
Pyrimethamine Blood levels | Weekly (1-18 weeks)
Pyrimethamine efficacy | 6 months
  Measurement of GM2 in blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Joe T Clarke, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada